CLINICAL TRIAL: NCT04647747
Title: Silent Hypoxia and Awake Proning in COVID-19 Patients: Home Monitoring and Self-Reporting
Brief Title: Silent Hypoxia and Awake Proning in COVID-19 Patients
Acronym: SHYCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Hans Joakim Myklebust-Hansen, Konstituert Overlege, Akuttseksjonen, Ostfold Hospital Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHYCOV2020
Record Dates: First submitted 2020-11-27; First posted 2020-12-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Covid19; Hypoxemia
Keywords: Silent Hypoxia; Lung Physiotherapy; Home Monitoring
MeSH Terms: conditions — COVID-19; Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self measurement of peripheral saturation (Other): Participant will be equipped with a pulse oximeter and perform saturation measurements.
  Interventions: Other: Self measurement with pulse oximeter

INTERVENTIONS:
Other: Self measurement with pulse oximeter — Participant will measure peripheral saturation at home, conduct physiotherapy if desaturation occurs, and contact hospital if desatuation persists
  Other Names: Lung physiotherapy

SUMMARY:
The Investigators want to examine patients infected with SARS-CoV-2 for the phenomenon "Silent Hypoxia", which is clinically significant hypoxia without corresponding degree of dyspnea. The patient population is infected individuals without any serious symptoms and is at home. The participants will be equipped with a pulse oximeter and a PEF-measurement device. Four times daily the participants will register saturation, degree of dyspnea and PEF. If the participants experience desaturation or increasing dyspnea, physiotherapy is to be performed, and if that doesn't relieve symptoms or increase oxygen saturation, the hospital should be contacted for admission. The first part of this study is a feasibility study, and if found feasible, the investigators will expand the study to more participants.

ELIGIBILITY:
Inclusion Criteria:

* Non dyspneic (NRS =/< 1) patients with positive SARS-CoV-2 test
* Age 18 - 80 years
* Patients managed at home
* Inclusion within 72 hours from positive test

Exclusion Criteria:

* Chronic hypoxia (SpO2 < 93 %) and/or first measured SpO2 < 93 %
* Admitted to hospital for COVID-19 prior to inclusion
* Unable to perform pulse oximetry
* Unable to perform physiotherapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of patients who manage to perform daily measurements of SpO2 | January 30, 2021
Incidence rate of silent hypoxia in non-hospitalized COVID-19 | January 30, 2021
Association between silent hypoxia and other subjective and objective measurements of disease severity | January 30, 2021

SECONDARY OUTCOMES:
Effect of a self-managed physiotherapy program on alleviating hypoxia | January 30, 2021
Rate of persistent silent hypoxia episode per patients | January 30, 2021
Rate of silent hypoxia episode per patients | January 30, 2021
Rate of hospital admission and ICU admission | January 30, 2021
Incidence of thromboembolic event in outpatients diagnosed with COVID-19 | January 30, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Ostfold Hospital, Sarpsborg, Grålum, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myklebust-Hansen HJ, Hasvik E, Solyga VM, Ghanima W. The feasibility of self-performing measurements of peripheral oxygen saturation and respiratory exercises in home-isolated COVID-19 patients-a single-arm prospective trial. Pilot Feasibility Stud. 2023 Dec 2;9(1):195. doi: 10.1186/s40814-023-01415-x. PMID 38042811